CLINICAL TRIAL: NCT00138957
Title: Laparoscopic Parastomal Hernia Repair Using an Innovative Composite Polypropylene Mesh - A Prospective Study
Brief Title: Study of a New Laparoscopic Technique for Parastomal Hernia Repair With Mesh
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: too few patients included
Sponsor: University Hospital, Gentofte, Copenhagen (Other)
Collaborators: Ethicon, Inc. (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: KA05102m
Record Dates: First submitted 2005-08-29; First posted 2005-08-30 (Estimated); Last update posted 2008-07-11 (Estimated); Status verified 2008-07

CONDITIONS: Hernia; Abdominal Hernia
Keywords: Laparoscopic parastomal hernia repair; Intraperitoneally; Mesh; Quality of life; Postoperative pain; Recurrence
MeSH Terms: conditions — Hernia; Hernia, Abdominal; Pain, Postoperative; Recurrence | interventions — Melanocyte-Stimulating Hormones

INTERVENTIONS:
Procedure: Laparoscopic parastomal hernia repair with mesh

SUMMARY:
The purpose of the study is to evaluate a new laparoscopic technique for parastomal hernia repair using an intraperitoneally placed Proceed mesh, looking at postoperative complications, recurrence rate and postoperative pain and quality of life.

DETAILED DESCRIPTION:
Parastomal hernia affects up to 50% of all patients following formation of a stoma, most often in patients with a colostomy. About 20% of the patients need surgical correction of their parastomal hernia. Symptoms associated with parastomal hernias goes from mild physical (pain) and cosmetic discomfort to life threatening conditions with obstruction, strangulation and perforation. Parastomal hernias have big socioeconomic consequences and remain a considerable clinical problem.

The surgical treatment of parastomal hernias is controversial. The best way to treat it is to restore the continuity of the intestine, but in permanent stomas, this is not an option. Many surgical techniques have been described when intervention is required, but the results are unacceptable. The traditional open techniques are local simple suturing of the fascia defect, stoma relocation, or repair with a prosthetic material either intraperitoneally or extraperitoneally (subfascial or onlay). Overall, the results of all methods are poor with high recurrence rates and high morbidity and mortality. Mesh repair has the lowest recurrence rate (0-39%) and stoma relocation and simple suture has reported recurrence rates on 0-76% and 46-100%, respectively. Laparoscopic repair of parastomal hernias with a prosthetic mesh inserted intraperitoneally is a new method described in a few small series. The results so far are encouraging, but the follow-up period is short.

Looking at the disappointing results from the traditional open techniques in the treatment of parastomal hernias together with the enormous success in laparoscopic ventral hernia repair and laparoscopy overall, we believe that laparoscopic parastomal hernia repair with mesh will be an effective treatment option in the future. Therefore, we find it interesting to investigate the technique in a prospective study

ELIGIBILITY:
Inclusion Criteria:

* Age 18 - 80 years
* Indication for laparoscopic parastomal hernia repair in general anaesthesia.
* Danish speaking
* ASA group I-III
* No remaining malignancy after former primary radical operation for colorectal cancer

Exclusion Criteria:

* Former operation (open/lap) for parastomal hernia with insertion of mesh, or other mesh operation in the area of herniation
* Incarcerated hernia (acute operation)
* History of abuse or permanent morphine use
* Expected bad compliance
* Current systemic steroid use or other immuno-suppressive treatment
* HIV-positive, pregnant or breast feeding
* Medical conditions contraindicating general anaesthesia
* Simultaneous operation for other ventral, inguinal or umbilical hernia
* Epidural or spinal anaesthesia
* Conversion to open procedure

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2005-09; Study Completion 2007-12 (Estimated)

PRIMARY OUTCOMES:
Recurrence of parastomal hernia after 6 months (ultrasound and clinical)
Postoperative pain (Visual Analog Scale, VAS 0-100, Verbal Rating Scale, VRS 0-3)
Stricture of stoma (Bougie, mm)
Quality of life (SF-36 and Ostomy Adjustment Scale (OAS))
General well-being (VAS 0-100)
Postoperative ileus/paralysis > 24 hours
Patient's satisfaction (VAS 0-100)
Bandage problems (VRS 0-3)

SECONDARY OUTCOMES:
Medical and surgical complications

CONTACTS AND LOCATIONS:
Overall Officials: Jacob Rosenberg, Prof, MD, Principal Investigator — Gentofte University Hospital, Dept. of Surgery